CLINICAL TRIAL: NCT02508766
Title: EFFECT OF MANUAL PLANTAR STIMULATION ON STATIC AND DYNAMIC POSTURAL CONTROL IN YOUNG HEALTHY SUBJECTS
Brief Title: Effect of Stimulating Plant on the Balance in Young Healthy
Acronym: Effplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ID010
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Postural Control; Plantar Stimulation; Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plantar stimulation (Experimental): The manipulation was performed with the subject in the supine position. The intervention lasted ten minutes and consisted of four stages: 5 glide pressures focused on each interdigital space, that lasted 10 seconds in duration, 5 compression-decompression of each metatarsophalangeal joint, 5 glide pressures applied for 5 seconds each, on the region of metatarsal heads, 5 static pressures applied for 10 seconds each, focused on four points of the sole.
  Interventions: Procedure: Plantar stimulation
- Control group (No Intervention): Volunteers received no intervention. They just sat there for 20 minutes before being evaluated.

INTERVENTIONS:
Procedure: Plantar stimulation — The manipulation was performed with the subject in the supine position. The intervention lasted ten minutes and consisted of four stages: 5 glide pressures focused on each interdigital space, that lasted 10 seconds in duration, 5 compression-decompression of each metatarsophalangeal joint, 5 glide pressures applied for 5 seconds each, on the region of metatarsal heads, 5 static pressures applied for 10 seconds each, focused on four points of the sole.
  Arms: Plantar stimulation

SUMMARY:
The primary purpose of this study was to examine the immediate effect of manual stimulation on the foot plant in static and dynamic balance in young healthy subjects. In addition, the secondary objectives of this study were: 1) to identify whether manual stimulation of the foot plant in healthy young subjects, carried out with an easily reproducible protocol with 10 minutes duration, improves static balance, measured with Unipedal Stance Test; 2) to assess whether, manual stimulation of the foot plant in healthy young subjects, carried out with an easily reproducible protocol with 10 minutes duration, improves dynamic balance test, measured with Star Excursion Balance Test.

DETAILED DESCRIPTION:
Methods Participants Participants from the University of Valencia (Spain) were asked to volunteer to participate in this study. Patients were included if they were university students and were able and willing to complete the protocol. Participants were excluded if they were ≥40 years-old or had a known musculoskeletal lower extremity injury (eg, postoperative conditions, musculotendinous or ligamentous problems), previous history of neurological problems, balance disorders (eg, vestibular or visual problems) or did some type of physical activity programme where balance exercises were performed.

Study design We conducted a randomized single-blind controlled study investigation. A non-stratified randomization list was generated and held centrally in sealed envelopes. Therefore, participants were randomly assigned to an experimental group, who received a plantar stimulation on the right foot, or to a control group, which did not receive any intervention.

Intervention Plantar stimulation In addition, a plantar stimulation directed at the plantar surface of the dominant foot was performed by an experienced physiotherapist, as described below. Participants performed one practice trial of plantar stimulation prior to performance. The manipulation was performed with the subject in the supine position. The intervention lasted ten minutes and consisted of four stages: 5 glide pressures focused on each interdigital space and on the internal longitudinal arch of the foot in a caudal direction, that lasted 10 seconds in duration, (2) 5 compression-decompression of each metatarsophalangeal joint, until a slight tension was perceived by the researcher at the joint, (3) 5 glide pressures applied for 5 seconds each, on the region of metatarsal heads, and (4) 5 static pressures applied for 10 seconds each, focused on four points of the sole: the head of the first and the fifth metatarsal head, the heel and the medial side of the midfoot (Figure 3). Duration of pressures was assessed by using an on-line metronome. Furthermore, all pressures, both static and glide, were measured by a strength dynamometer and the mean force of pressure was 48N. After the stimulation, given to the negative effects of the sudden standing-up on several study results, participants stood quietly for 20 seconds before balance tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they were healthy university students and were able and willing to complete the protocol

Exclusion Criteria:

* Had a known musculoskeletal lower extremity injury (eg, postoperative conditions, musculotendinous or ligamentous problems).
* Previous history of neurological problems.
* Balance disorders (eg, vestibular or visual problems).
* Did some type of physical activity programme where balance exercises were performed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements (the measure is a composite) | 1 day
  * Height (cm)
  * Mass (kg). Body mass index was calculated from height and mass data (kg/m2).
  * Bilateral leg length measures (cm). On a plinth with participant in supine, leg length was assessed using a standard tape measure. The distance between the anterior superior iliac spine and the most distal portion of the medial malleolus of the same leg was measured. Both legs were evaluated.

SECONDARY OUTCOMES:
Static postural control testing: Unipedal Stance Test | 1 day
  Static balance was assessed using the UPST. Firstly, participants were asked to focus on a spot on the wall at eye level in front of them. Then, they had to cross their arms over the chest and close their eyes. Afterwards, subjects had to undergo the test barefoot standing on one leg on a stable surface, while maintaining balance for as long as possible up to a 45 second period. A stopwatch was used to determine the elapsed time the student was able to maintain unipedal stance up to a maximum of 45 seconds. The trial was disregarded and repeated when participants (1) touched the floor or moved the free foot from the standing limb, (2) uncrossed their arms, (3) moved the standing foot to maintain his balance or (4) opened eyes. Finally, subjects then completed 3 test trials, sitting in a chair to rest for 5 minutes. The average score of the amount of time of three trials was recorded.
Dynamic postural control testing: Star Excursion Balance Test. | 1 day
  Consists of 8 directions, whilst several studies have confirmed the utility of a reduced version of the test using the anterior (ANT), posteromedial (PM) and posterolateral (PL) reaching directions. Participants were required to reach with the free limb for maximal distance in each of three directions and then lightly touch one line, while maintaining his/her balance and without using the free limb for support. Then, 3 trials in each direction for each limb were performed. Visual cues (objects on the floor, people not participating in the study, etc.) were avoided, in order to reduce visual and auditory influences. The trial was repeated when (1) the reach limb touched heavily at the floor, in order to maintain balance or to get any support, (2) moved the stance foot from the grid, (3) failed to return the reach foot to the starting position, or (4) subject's hands did not remain on his/her hips.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, PhD, Principal Investigator — Faculty of Physiotherapy

REFERENCES:
- [Result] Hatton AL, Dixon J, Rome K, Newton JL, Martin DJ. Altering gait by way of stimulation of the plantar surface of the foot: the immediate effect of wearing textured insoles in older fallers. J Foot Ankle Res. 2012 Apr 30;5:11. doi: 10.1186/1757-1146-5-11. PMID 22546376
- [Result] Hurvitz EA, Richardson JK, Werner RA, Ruhl AM, Dixon MR. Unipedal stance testing as an indicator of fall risk among older outpatients. Arch Phys Med Rehabil. 2000 May;81(5):587-91. doi: 10.1016/s0003-9993(00)90039-x. PMID 10807096
- [Result] Muir J, Judex S, Qin YX, Rubin C. Postural instability caused by extended bed rest is alleviated by brief daily exposure to low magnitude mechanical signals. Gait Posture. 2011 Mar;33(3):429-35. doi: 10.1016/j.gaitpost.2010.12.019. Epub 2011 Jan 26. PMID 21273076